CLINICAL TRIAL: NCT04383327
Title: Effectiveness and Implementation of an Early Childhood School-Based Mental Health Intervention in Low-Resource Communities
Brief Title: School-Based Mental Health Effectiveness Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20-00117
Record Dates: First submitted 2020-04-16; First posted 2020-05-12 (Actual); Results first posted 2025-08-08 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-07

CONDITIONS: Child Development

STUDY DESIGN:
Intervention Model Description: A cluster randomized controlled trial (cRCT), single blind and mixed-methods design will be applied
Who Masked: Outcomes Assessor
Masking Description: Research staff performing outcome assessment will be blind to the study conditions.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ParentCorps-Professional Development (PD) (Experimental): n = 6 Schools in Kampala, Uganda (Urban) - 89 Teachers, 325 Parent-Child Pairs
  + n = 10 Schools in Hoima, Uganda (Rural) - 98 Teachers, 344 Parent-Child Pairs
  Interventions: Behavioral: ParentCorps-Professional Development (PD)
- ParentCorps-Professional Development (PD) + T-Wellness (Experimental): n = 6 Schools in Kampala, Uganda (Urban) - 77 Teachers, 300 Parent-Child Pairs
  + n = 10 Schools in Hoima, Uganda (Rural) - 80 Teachers, 329 Parent-Child Pairs
  Interventions: Behavioral: ParentCorps-Professional Development (PD); Behavioral: T-Wellness
- Control (No Intervention): n = 6 Schools in Kampala, Uganda (Urban) - 73 Teachers, 316 Parent-Child Pairs
  + n = 9 Schools in Hoima, Uganda (Rural) - 92 Teachers, 321 Parent-Child Pairs

INTERVENTIONS:
Behavioral: ParentCorps-Professional Development (PD) — Multi-component school-based intervention that promotes early childhood mental health and development. Teachers (pre-primary to 4th grade) will participate in a 3-day ParentCorps-PD training during the school term. They will also receive 8 sessions (8 hours) of face-to-face group-based coaching during after the training. Coaching sessions are to help teachers apply EBI strategies in their classrooms, engage families, and develop competencies.
  Arms: ParentCorps-Professional Development (PD); ParentCorps-Professional Development (PD) + T-Wellness
Behavioral: T-Wellness — A brief teacher stress management psychoeducation package, adapted from EBIs including one-day workshop for common stress management and stress management, and three follow-up group support sessions (3 additional monthly 1-hr wellness sessions for teachers as a group that were integrated into the 3 of the 8 PD coaching sessions. A total 3 hours of coaching were included.
  Arms: ParentCorps-Professional Development (PD) + T-Wellness

SUMMARY:
This study involves efforts to advance the science of prevention in early childhood mental health in low-resource communities. Investigators will assess the effectiveness, practical implementation strategies, and underlying mechanisms of the evidence-based intervention, ParentCorps-Professional Development, in urban and rural Uganda. Two implementation approaches, with and without the teacher stress management package, T-Wellness, will be compared for efficacy.

DETAILED DESCRIPTION:
Promoting child mental health in low-resource or low-income country settings faces numerous challenges in global health research. Although efforts have been made to improve mental health interventions and services for young children, evidence-based interventions (EBIs) for children in low-and middle-income countries (LMICs) are limited. Most mental health EBIs in LMICs have not been scaled widely, and do not focus on early childhood. Mechanisms of action and effectiveness are not well understood. Additionally, most EBIs in LMICs rely on community health workers (CHWs) or a task-shifting approach of implementation because of resource barriers and shortage of mental health professionals (MHPs). However, challenges related to task-shifting (e.g., CHW stress and job burnout) have rarely been studied. For task-shifting to be successful, strategies to overcome challenges faced by CHWs and understanding mechanisms to conduct effective task-shifting are paramount. The overall goal of this study is to address these EBI effectiveness and implementation knowledge gaps by providing a preventive EBI (ParentCorps-Professional Development; PD) that utilizes a task-shifting and a scalable implementation model to promote early childhood students' mental health in a LMIC-Uganda. PD is a school-based EBI and preventive mental health service provision model that supports teachers and school personnel to apply EBI strategies to promote young children's mental health. The PD approach represents a task-shifting model of mental healthcare by shifting mental health preventive duties from professionals to teachers to optimize school children's mental health. Therefore, teachers are considered as CHWs. This study examines impacts and cost-effectiveness of the EBI/PD on teachers and students, as well as examines underlying mechanisms (or theories of change) that contribute to intervention effect. In addition, considering most Ugandan teachers (or CHWs) experience occupational stress that threatens PD uptake, effectiveness, and sustainment, this study will also test a teacher stress management package (T-Wellness, adapted from EBIs) as an enhancement to PD. This study will investigate whether PD + T-Wellness (PDT) is more effective for CHWs/teachers than PD alone.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria:

1. The inclusion criteria for the school staff (teachers, head teachers) are: they must be in the recruited study schools and teaching in Pre-Primary to Primary 4 classrooms or holding the head teachers/administration leadership position in school. The inclusion criteria for Parent Leaders are: they must be at least 18 years old and have served as a Parent-Teacher-Association member or Parent Leader in the school for at least 1 year.
2. The inclusion criteria for the PD/PDT program implementers are: they must have current employment with eligible partners (i.e., medical/mental health institutions, Teacher Training Colleges), with professional experiences in teacher training or mental health training.
3. The inclusion criteria for parents are: caregivers must be at least 18 years old, their children must be enrolled in Pre-Primary or Primary 1 to 4 classes (or between 3 to 10 years old) in the recruited schools, and willing to have their child to be assessed by research staff. Parents and children will have diverse characteristics (e.g., randomly selected from school student lists). About 10% families will be randomly selected from the student lists. The proposed study will be open to both men and women caregivers

Exclusion Criteria

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Evidence of psychopathology or cognitive impairment severe enough to preclude giving consent, or completing the survey instruments or the focus group of the study.
2. Minors (age <18) will also be excluded. Additional criteria should be included as appropriate for the study design and risk.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2444 (Actual)
Dates: Start 2021-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keng-Yen Huang, MD, MPH, Principal Investigator — NYU Langone Health
Locations (2):
- Uganda (2):
  - Hoima School, Hoima
  - Kampala School, Kampala

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research datasets (defined below) will be shared via the National Databased of Clinical Trials (NDCT) related to Mental Illness. The proposed cluster RCT study will be carried out in Uganda. It will collect data on 540 school staff (i.e., teachers), and 1,980 parent-child pairs from 36 schools. Child and teacher/school effectiveness outcome data and demographic data collected from teachers, schools, and families across all three assessment time points will be released for sharing. In addition, implementation context data will also be released. These data will be share via the NDCT related to Mental Illness. Implementation fidelity data will not be shared through NDCT, but can be requested from the PI Keng-Yen Huang directly beginning 9 months following article publication or at the end of the study.
Supporting Information: Study Protocol, SAP
Time Frame: Analyzed data file and final trial data will be share at the end of the study via the National Databased of Clinical Trials (NDCT) related to Mental Illness (the NIMH recommended format). There will be no end date for data sharing.
Access Criteria: Requests should be directed to PI Keng-Yen Huang at huangk01@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Derived] Huang KY, Nakigudde J, Kisakye EN, Sentongo H, Dennis-Tiwary TA, Tozan Y, Park H, Brotman LM. Advancing scalability and impacts of a teacher training program for promoting child mental health in Ugandan primary schools: protocol for a hybrid-type II effectiveness-implementation cluster randomized trial. Int J Ment Health Syst. 2022 Jun 20;16(1):28. doi: 10.1186/s13033-022-00538-7. PMID 35718782

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: While parents + children were enrolled as dyads, only the parent participants provided consent. The participant flow information provides the total number of parents AND children. The baseline characteristic information provides data on parents only, as only parents had baseline characteristic data collected. Further, all child-related assessments were completed by the parent participants.
Units Other Than Participants: Schools
Groups:
- ParentCorps-Professional Development (PD) - Parent + Child: Urban: Parents + Children assigned to the PD-only group in an urban setting.
- ParentCorps-Professional Development (PD) - Teachers: Urban: Teachers assigned to the PD-only group in an urban setting.
- ParentCorps-Professional Development (PD) + T-Wellness - Parent + Child: Urban: Parents + Children assigned to the PD+T wellness group in an urban setting.
- ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban: Teachers assigned to the PD+T wellness group in an urban setting.
- Control - Parent + Child: Urban: Parents + Children assigned to the control group in an urban setting.
- Control - Teacher: Urban: Teachers assigned to the control group in an urban setting.
- ParentCorps-Professional Development (PD) - Parent + Child: Rural: Parents + Children assigned to the PD-only group in a rural setting.
- ParentCorps-Professional Development (PD) - Teachers: Rural: Teachers assigned to the PD-only group in a rural setting.
- ParentCorps-Professional Development (PD) + T-Wellness - Parent + Child: Rural: Parents + Children assigned to the PD+T wellness group in a rural setting.
- ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Rural: Teachers assigned to the PD+T wellness group in a rural setting.
- Control - Parent + Child: Rural: Parents + Children assigned to the control group in a rural setting.
- Control - Teacher: Rural: Teachers assigned to the control group in a rural setting.
Period: Overall Study
Arm/Group | ParentCorps-Professional Development (PD) - Parent + Child: Urban | ParentCorps-Professional Development (PD) - Teachers: Urban | ParentCorps-Professional Development (PD) + T-Wellness - Parent + Child: Urban | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban | Control - Parent + Child: Urban | Control - Teacher: Urban | ParentCorps-Professional Development (PD) - Parent + Child: Rural | ParentCorps-Professional Development (PD) - Teachers: Rural | ParentCorps-Professional Development (PD) + T-Wellness - Parent + Child: Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Rural | Control - Parent + Child: Rural | Control - Teacher: Rural
Started | 650; 6 Schools (The number of participants represents the total number of parents + children; n = 325 dyads started the study.) | 89; 6 Schools | 600; 6 Schools (The number of participants represents the total number of parents + children; n = 300 dyads started the study.) | 77; 6 Schools | 632; 6 Schools (The number of participants represents the total number of parents + children; n = 316 dyads started the study.) | 73; 6 Schools | 688; 10 Schools (The number of participants represents the total number of parents + children; n = 344 dyads started the study.) | 98; 10 Schools | 658; 10 Schools (The number of participants represents the total number of parents + children; n = 329 dyads started the study.) | 80; 10 Schools | 642; 9 Schools (The number of participants represents the total number of parents + children; n = 321 dyads started the study.) | 92; 9 Schools
Completed | 538; 6 Schools (The number of participants represents the total number of parents + children; n = 269 dyads completed the study.) | 75; 6 Schools | 522; 6 Schools (The number of participants represents the total number of parents + children; n = 261 dyads completed the study.) | 64; 6 Schools | 522; 6 Schools (The number of participants represents the total number of parents + children; n = 261 dyads completed the study.) | 60; 6 Schools | 614; 10 Schools (The number of participants represents the total number of parents + children; n = 307 dyads completed the study.) | 85; 10 Schools | 580; 10 Schools (The number of participants represents the total number of parents + children; n = 290 dyads completed the study.) | 70; 10 Schools | 482; 9 Schools (The number of participants represents the total number of parents + children; n = 241 dyads completed the study.) | 79; 9 Schools
Not Completed | 112; 0 Schools | 14; 0 Schools | 78; 0 Schools | 13; 0 Schools | 110; 0 Schools | 13; 0 Schools | 74; 0 Schools | 13; 0 Schools | 78; 0 Schools | 10; 0 Schools | 160; 0 Schools | 13; 0 Schools
Not completed — Lost to Follow-up | 112 | 14 | 78 | 13 | 110 | 13 | 74 | 13 | 78 | 10 | 160 | 13

BASELINE CHARACTERISTICS:
Population: Note that only parent participants in the parent + child dyads were consented and had baseline characteristic data collected.
Groups:
- ParentCorps-Professional Development (PD) - Parents Urban: Parents of school children assigned to the PD-only group in an urban setting.
- ParentCorps-Professional Development (PD) + T-Wellness - Parents: Urban: Parents of school children assigned to the PD+T wellness group in an urban setting.
- Control - Parents: Urban: Parents of school children assigned to the control group in an urban setting.
- ParentCorps-Professional Development (PD) - Parents: Rural: Parents of school children assigned to the PD-only group in a rural setting.
- ParentCorps-Professional Development (PD) + T-Wellness - Parents: Rural: Parents of school children assigned to the PD+T wellness group in a rural setting.
- Control - Parents: Rural: Parents of school children assigned to the control group in a rural setting.
- Total: Total of all reporting groups
Arm/Group | ParentCorps-Professional Development (PD) - Parents Urban | ParentCorps-Professional Development (PD) - Teachers: Urban | ParentCorps-Professional Development (PD) + T-Wellness - Parents: Urban | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban | Control - Parents: Urban | Control - Teacher: Urban | ParentCorps-Professional Development (PD) - Parents: Rural | ParentCorps-Professional Development (PD) - Teachers: Rural | ParentCorps-Professional Development (PD) + T-Wellness - Parents: Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Rural | Control - Parents: Rural | Control - Teacher: Rural | Total
Number analyzed (Participants) | 325 | 89 | 300 | 77 | 316 | 73 | 344 | 98 | 329 | 80 | 321 | 92 | 2444
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.04 (9.65) | 40.9 (11.8) | 36.54 (10.17) | 40.2 (12.3) | 35.83 (8.86) | 42.7 (11.3) | 38.07 (10.63) | 40.8 (9.7) | 38.05 (9.46) | 40.8 (11.8) | 38.33 (11.49) | 38.4 (9.9) | 38.88 (10.59)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 245 | 68 | 250 | 49 | 237 | 50 | 232 | 74 | 239 | 64 | 211 | 63 | 1782
  Male | 80 | 21 | 50 | 28 | 79 | 23 | 112 | 24 | 90 | 16 | 110 | 29 | 662
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 325 | 89 | 300 | 77 | 316 | 73 | 344 | 98 | 329 | 80 | 321 | 92 | 2444
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 325 | 89 | 300 | 77 | 316 | 73 | 344 | 98 | 329 | 80 | 321 | 92 | 2444
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Uganda | 325 | 89 | 300 | 77 | 316 | 73 | 344 | 98 | 329 | 80 | 321 | 92 | 2444

OUTCOME MEASURES:

1. Primary Outcome: Teacher Knowledge of Evidence-Based Practice (Knowledge Score)
Description: Teachers will complete a 10-item quiz assessing EBI knowledge. The total score is the number of correct responses and ranges from 0-100; higher scores indicate greater knowledge.
Time Frame: Baseline
Population: All teacher participants were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ParentCorps-Professional Development (PD) - Teachers: Urban and Rural: Teachers assigned to the PD-only group.
- ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural: Teachers assigned to the PD+T wellness group.
- Control - Teacher: Urban and Rural: Teachers assigned to the control group.
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 187 | 157 | 165
score on a scale | 36.68 (14.46) | 36.41 (13.96) | 35.18 (11.75)

2. Primary Outcome: Teacher Knowledge of Evidence-Based Practice (Knowledge Score)
Description: as for outcome 1
Time Frame: Month 6
Population: Mean values are reported based on the raw data using cases with the follow up data. However, effectiveness outcome analysis were conducted based on the entire sample using imputated data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 142 | 126 | 123
score on a scale | 41.91 (15.85) | 45.12 (14.12) | 36.75 (13.64)

3. Primary Outcome: Teacher EBI Practice Score-Emotion Support Strategies Use
Description: The Emotion Socialization Scale assesses teachers' practice in supporting students' management of negative emotions. Each of the scale items (6 items) are rated on a scale from 1 to 5. The total score is the average of responses and ranges from 1-5; lower scores indicate lower adherence to EBI practice.
Time Frame: Baseline
Population: All teacher participants were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 187 | 157 | 165
score on a scale | 3.92 (0.79) | 3.91 (0.74) | 3.77 (0.83)

4. Primary Outcome: Teacher EBI Practice Score-Emotion Support Strategies Use
Description: as for outcome 3
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 142 | 126 | 123
score on a scale | 3.83 (0.80) | 4.06 (0.71) | 3.74 (0.81)

5. Primary Outcome: Teacher EBI Practice Score-Emotion Support Strategies Use
Description: as for outcome 3
Time Frame: Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 149 | 114 | 118
score on a scale | 4.14 (0.75) | 4.19 (0.63) | 3.98 (0.77)

6. Primary Outcome: Teacher Stress Score
Description: Teachers complete a 5-item assessment of stress over the past month. Each item is rated on a scale from 1 to 4. The total score is the average of responses and ranges from 1-4. Higher scores indicate greater stress.
Time Frame: Baseline
Population: All teacher participants were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 187 | 157 | 165
score on a scale | 1.98 (0.63) | 2.05 (0.66) | 2.07 (0.58)

7. Primary Outcome: Teacher Stress Score
Description: as for outcome 6
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 142 | 126 | 123
score on a scale | 1.79 (0.63) | 1.77 (0.49) | 1.93 (0.6)

8. Primary Outcome: Teacher Stress Score
Description: as for outcome 6
Time Frame: Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 149 | 114 | 118
score on a scale | 1.84 (0.75) | 1.83 (0.68) | 1.83 (0.58)

9. Primary Outcome: Child's Emotion Regulation Score
Description: Parents answer 6 questions about their child's emotion regulation behavior over the past 7 days. Each item is rated on a Likert scale from 0 (not at all) to 4 (very well). The total score ranges from 0 to 4; higher scores indicate greater emotion regulation.
Time Frame: Baseline
Population: All parent participants' data are analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- ParentCorps-Professional Development (PD) - Parents: Urban and Rural: Parents assigned to the PD-only group.
- ParentCorps-Professional Development (PD) + T-Wellness - Parents: Urban and Rural: Parents assigned to the PD+T wellness group.
- Control - Parents: Urban and Rural: Parents assigned to the control group.
Arm/Group | ParentCorps-Professional Development (PD) - Parents: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Parents: Urban and Rural | Control - Parents: Urban and Rural
Number analyzed (Participants) | 669 | 629 | 637
score on a scale | 2.33 (0.77) | 2.42 (0.73) | 2.39 (0.75)

10. Primary Outcome: Child's Emotion Regulation Score
Description: as for outcome 9
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Parents: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Parents: Urban and Rural | Control - Parents: Urban and Rural
Number analyzed (Participants) | 421 | 441 | 361
score on a scale | 2.71 (0.65) | 2.75 (0.68) | 2.58 (0.7)

11. Primary Outcome: Child's Emotion Regulation Score
Description: as for outcome 9
Time Frame: Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Parents: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Parents: Urban and Rural | Control - Parents: Urban and Rural
Number analyzed (Participants) | 515 | 474 | 446
score on a scale | 2.56 (0.64) | 2.47 (0.63) | 2.53 (0.64)

12. Secondary Outcome: Teacher Mental Health
Description: Teachers complete Kessler Psychological Distress Scale (K10), which assesses anxiety and depressive symptoms that teacher experiencing over the past month. Each item is rated on a scale from 0 to 4. The total score is the sum of responses and ranges from 0 to 40, where higher scores indicate greater psychological distress.
Time Frame: Baseline
Population: All teacher participants were analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 187 | 157 | 165
score on a scale | 20.74 (5.62) | 21.54 (6.68) | 20.55 (5.81)

13. Secondary Outcome: Teacher Mental Health
Description: as for outcome 12
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 142 | 126 | 123
score on a scale | 18.55 (6.01) | 18.84 (5.17) | 19.77 (6.24)

14. Secondary Outcome: Teacher Mental Health
Description: as for outcome 12
Time Frame: Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Teachers: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Teachers: Urban and Rural | Control - Teacher: Urban and Rural
Number analyzed (Participants) | 149 | 114 | 118
score on a scale | 18.79 (5.96) | 18.82 (5.55) | 19.32 (5.94)

15. Secondary Outcome: Child Mental Health- Conduct Problem
Description: Conduct problem items (5 items) from the Strengths and Difficulties Questionnaire (SDQ) are rated by parents, which assesses child's conduct and non-compliant behaviors over the last six months. Each item is rated on a Likert scale from 0 (not true) to 2 (certainly true). The total score is the sum of responses and ranges from 0-10; higher scores indicate greater difficulties.
Time Frame: Baseline
Population: All parent participants are analyzed.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Parents: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Parents: Urban and Rural | Control - Parents: Urban and Rural
Number analyzed (Participants) | 669 | 629 | 637
score on a scale | 2.39 (2.05) | 2.41 (1.98) | 2.44 (2.09)

16. Secondary Outcome: Child Mental Health- Conduct Problem
Description: as for outcome 15
Time Frame: Month 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Parents: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Parents: Urban and Rural | Control - Parents: Urban and Rural
Number analyzed (Participants) | 421 | 441 | 361
score on a scale | 1.96 (1.81) | 2.23 (1.90) | 2.13 (1.95)

17. Secondary Outcome: Child Mental Health- Conduct Problem
Description: as for outcome 15
Time Frame: Month 18
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | ParentCorps-Professional Development (PD) - Parents: Urban and Rural | ParentCorps-Professional Development (PD) + T-Wellness - Parents: Urban and Rural | Control - Parents: Urban and Rural
Number analyzed (Participants) | 515 | 474 | 446
score on a scale | 1.76 (1.76) | 1.71 (1.69) | 1.77 (1.64)

ADVERSE EVENTS:
Time Frame: Two years.
Groups:
- ParentCorps-Professional Development (PD): n = 6 Schools in Kampala, Uganda (Urban) - 89 Teachers, 325 Parent-Child Pairs
  + n = 10 Schools in Hoima, Uganda (Rural) - 98 Teachers, 344 Parent-Child Pairs
  ParentCorps-Professional Development (PD): Multi-component school-based intervention that promotes early childhood mental health and development. Teachers (pre-primary to 4th grade) will participate in a 3-day ParentCorps-PD training during the school term. They will also receive 8 sessions (8 hours) of face-to-face group-based coaching during after the training. Coaching sessions are to help teachers apply EBI strategies in their classrooms, engage families, and develop competencies.
- ParentCorps-Professional Development (PD) + T-Wellness: n = 6 Schools in Kampala, Uganda (Urban) - 77 Teachers, 300 Parent-Child Pairs
  + n = 10 Schools in Hoima, Uganda (Rural) - 80 Teachers, 329 Parent-Child Pairs
  ParentCorps-Professional Development (PD): Multi-component school-based intervention that promotes early childhood mental health and development. Teachers (pre-primary to 4th grade) will participate in a 3-day ParentCorps-PD training during the school term. They will also receive 8 sessions (8 hours) of face-to-face group-based coaching during after the training. Coaching sessions are to help teachers apply EBI strategies in their classrooms, engage families, and develop competencies.
  T-Wellness: A brief teacher stress management psychoeducation package, adapted from EBIs including one-day workshop for common stress management and stress management, and three follow-up group support sessions (3 additional monthly 1-hr wellness sessions for teachers as a group that were integrated into the 3 of the 8 PD coaching sessions. A total 3 hours of coaching were included.
Arm/Group | ParentCorps-Professional Development (PD) | ParentCorps-Professional Development (PD) + T-Wellness | Control
All-Cause Mortality (participants affected / at risk) | 0/1525 | 0/1415 | 0/1439
Serious Adverse Events (participants affected / at risk) | 0/1525 | 0/1415 | 0/1439
Other Adverse Events (participants affected / at risk) | 0/1525 | 0/1415 | 0/1439

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT04383327/Prot_SAP_000.pdf